CLINICAL TRIAL: NCT04758104
Title: Assessment of the Efficacy of Stereotactic Intracavitary Instillation of 90Yttrium Colloid for Treatment of Cystic Lesions of the Brain: Open Label Individual Patient (OLIP) Study
Brief Title: Assessment of the Efficacy of Stereotactic Intracavitary Instillation of 90Yttrium Colloid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Clarke (Other)
Collaborators: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, David Clarke, Neurosurgeon, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1026510
Record Dates: First submitted 2021-02-05; First posted 2021-02-17 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Neuroepithelial Cyst
MeSH Terms: conditions — Colloid cysts of third ventricle | interventions — Yttrium-90

STUDY DESIGN:
Intervention Model Description: To estimate the efficacy of intracavitary application of 90Yttrium colloid for the treatment of an adult with a cystic tumor in the brain by a single neurosurgeon.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yttrium90 (Experimental): Intracystic application of yttrium90
  Interventions: Radiation: Yttrium90

INTERVENTIONS:
Radiation: Yttrium90 — Intracystic implantation of 90yttrium colloid

SUMMARY:
Neuroepithelial cysts are rare, representing less than 1% of the intracranial cysts. Neuroepithelial cysts, are benign and mostly asymptomatic. These cysts are lined by thin columnar or low cuboidal epithelium. The CSF-like contents of the cyst are due to secretion of the epithelial cyst wall. Although mostly asymptomatic, symptoms can occur when the cyst enlarges; the specific symptoms vary according to the size (mass effect) and location of the lesion. Radioactive phosphorus (32P) and 90yttrium colloid are isotopes that have been used. These are approved in the United States and Europe. 32P is not available in Canada. We want to use 90yttrium colloid. There is evidence in the scientific literature that treatment with 90yttrium colloid injected into the cyst is effective in preventing the cyst from growing, effective in causing the cyst to get smaller and in some cases the cyst disappears.

DETAILED DESCRIPTION:
In brief, a single patient has been identified as having a cystic tumor by diagnostic imaging and clinical expertise and based on standards of excellence in clinical care will be offered participation in the study for the intracystic implantation of 90yttrium colloid. This patient will be followed closely for 4 weeks following 90yttrium colloid treatment and then receive standard of care (http://neurosurgery.medicine.dal.ca).

ELIGIBILITY:
Inclusion criteria:

1. Cystic tumor
2. Required treatment
3. Adult over 17 years of age
4. Willingness to provide informed consent

Exclusion criteria

1. Solid tumor
2. Treatment not required
3. Child under 17 years of age
4. Not willing to provide informed consent

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-01-24 (Actual)

PRIMARY OUTCOMES:
Demonstration of intracavitary application of 90Yttrium colloid into a cystic tumor in the brain. | 1 MONTH
  90Yttrium colloid will be inserted into the cyst using neurosurgical techniques.
Shrinkage of cyst | 1 Month
  Intracystic application of 90Yttrium colloid will result in the shrinkage of the cyst.To estimate the efficacy of intracavitary application of 90Yttrium colloid for the treatment of an adult with a cystic tumor in the brain by a single neurosurgeon.

SECONDARY OUTCOMES:
PET-CT scan will be used to visualize the yttrium within the cyst. | 1 -4 days
  We will be evaluating the utility of positron emission tomography - computed tomography (PET-CT) in demonstrating that the distribution of 90yttrium colloid is confined to the cyst.

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No